CLINICAL TRIAL: NCT00841425
Title: Airway Responsiveness and Inflammation in Adolescent Elite Swimmers: a 3-Year Prospective Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Lars Pedersen (MD PhD), Respiratory and Allergy Research Unit, Bispebjerg Hospital, Copenhagen, Denmark
Other Study IDs: H-B-2009-012
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (serum, whole blood) Exhaled breath condensate Induced sputum

GROUPS / COHORTS (1):
- Swimmers

SUMMARY:
Previously the investigators have found that adolescent elite swimmers, who have been involved in competitive swimming for only a few years, have not developed respiratory symptoms, signs of airway inflammation or airway hyperresponsiveness exept for a slight increase in airway responsiveness to eucapnic voluntary hyperpnea. In the current study, the investigators will be doing a 3-year follow-up study on the swimmers studied previously.

DETAILED DESCRIPTION:
Even though studies suggest that elite sport can cause AHR and airway inflammation, more studies are needed to elucidate how and when AHR and airway inflammation develop; and there is a lack of follow-up studies. The present study will give us a chance to do a follow-up study to register changes in AHR and airway inflammation in athletes without any significant airway changes at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-19 years
* Part of the Danish National Swimming Association's talent program for young swimmers at the baseline study
* Informed consent

Exclusion Criteria:

* Upper respiratory tract infection in the previous 4 weeks (visits will be postponed)

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants were all elite swimmers and part of the Danish National Swimming Association's talent program for young swimmers at the baseline study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Airway responsiveness to eucapnic voluntary hyperpnea and methacholine | Three years

SECONDARY OUTCOMES:
Airway inflammation | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Pedersen, MD PhD, Principal Investigator — Respiratory and Allergy Research Unit, Bispebjerg Hospital
Locations (1):
- Respiratory and Allergy Research Unit, Department of Respiratory Medicine L, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Pedersen L, Lund TK, Barnes PJ, Kharitonov SA, Backer V. Airway responsiveness and inflammation in adolescent elite swimmers. J Allergy Clin Immunol. 2008 Aug;122(2):322-7, 327.e1. doi: 10.1016/j.jaci.2008.04.041. Epub 2008 Jun 12. PMID 18554704